CLINICAL TRIAL: NCT04085601
Title: A Phase 3, Randomized, Multicenter, Open-Label, Controlled Study to Evaluate the Efficacy and Safety of Pegcetacoplan in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: A Study to Evaluate the Efficacy and Safety of Pegcetacoplan in Patients With PNH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APL2-308
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Results first posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) excluding complement inhibitors (No Intervention)
- 1,080mg APL-2 administered subcutaneously twice weekly (Experimental)
  Interventions: Drug: APL-2

INTERVENTIONS:
Drug: APL-2 — Complement (C3) Inhibitor
  Arms: 1,080mg APL-2 administered subcutaneously twice weekly

SUMMARY:
Evaluation of the Efficacy and Safety of Pegcetacoplan in Patients with Paroxysmal Nocturnal Hemoglobinuria .

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old (inclusive).
* Have LDH ≥1.5 x ULN at the screening visit.
* Have PNH diagnosis, confirmed by high sensitivity flow cytometry (granulocyte or monocyte clone >10%).
* Have Hb less than the lower limit of normal (LLN) at the screening visit.
* Have ferritin greater than/equal to the LLN, or total iron binding capacity (TIBC) less than/equal to ULN at the screening visit, based on central laboratory reference ranges. If a subject is receiving iron supplements at screening, the Investigator must ensure that the subject's dose has been stable for 4 weeks prior to screening, and it must be maintained throughout the study. Subjects not receiving iron at screening must not start iron supplementation during the course of the study.
* Body mass index (BMI) ≤ 35 kg/m2 at the screening visit.
* Have a platelet count of >50,000/mm3 at the screening visit.
* Have an absolute neutrophil count >500/mm3 at the screening visit.

Exclusion Criteria:

* Treatment with any complement inhibitor (eg, eculizumab) within 3 months prior to screening.
* Hereditary complement deficiency.
* History of bone marrow transplantation.
* Concomitant use of any of the following medications is prohibited if not on a stable regimen for the time period indicated below prior to screening:

  * Erythropoietin or immunosuppressants for at least 8 weeks
  * Systemic corticosteroids for at least 4 weeks
  * Vitamin K antagonists (eg, warfarin) with a stable international normalized ratio (INR) for at least 4 weeks
  * Iron supplements, vitamin B12, or folic acid for at least 4 weeks
  * Low-molecular-weight heparin for at least 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- Colombia (2):
  - Julian Coronel Medical Center, Cali
  - Research Center of the Colombian Clinical Life Cancer Foundation, Medellín
- Hong Kong (3):
  - Queen Mary Hospital, Hong Kong
  - Princess Margaret Hospital, Kwai Chung
  - Prince and Wales Hospital, Shatin
- Malaysia (2):
  - Hospital Ampang, Ampang, Selangor
  - University Malaya Medical Centre, Kuala Lumpur
- Hospital Universitario Dr.Jose Eleuterio Gonzalez, Monterrey, Mexico
- Peru (3):
  - Hospital Cayetano Heredia, San Martín de Porres, Lima region
  - Hospital Cayetano Heredia, Jesús María, Lima
  - Hospital Nacional Dos de Mayo, Lima
- Philippines (6):
  - Baguio General Hospital, Benguet
  - Perpetual Succour Hospital, Cebu City
  - Mary Mediatrix Medical Center, Lipa City
  - Makati Medical Centre, Makati City
  - The Medical City, Pasig
  - St. Lukes Medical Centre, Quezon City
- Poland (3):
  - Independent Public Clinical Hospital, Lubin
  - Institute of Hematology and Transfusiology, Warsaw
  - EMC Medical Institute, Wroclaw
- Clinical Centre of Serbia, Belgrade, Serbia
- Singapore General Hospital (SGH), Singapore, Singapore
- Thailand (8):
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Hospital for Tropical disease, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagaring Hospital, Khon Kaen
  - Thammasat University Hospital, Pathum Thani
  - Songklanagaring Hospital, Songkhla

REFERENCES:
- [Derived] de Castro C, Kelly RJ, Griffin M, Patriquin CJ, Mulherin B, Hochsmann B, Selvaratnam V, Wong RSM, Hillmen P, Horneff R, Uchendu UO, Zhang Y, Surova E, Szamosi J, de Latour RP. Efficacy and Safety Maintained up to 3 Years in Adults with Paroxysmal Nocturnal Hemoglobinuria Receiving Pegcetacoplan. Adv Ther. 2025 Sep;42(9):4641-4658. doi: 10.1007/s12325-025-03310-8. Epub 2025 Jul 28. PMID 40720060
- [Derived] Panse J, Daguindau N, Okuyama S, Peffault de Latour R, Schafhausen P, Straetmans N, Al-Adhami M, Persson E, Wong RSM. Improvements in hematologic markers and decreases in fatigue with pegcetacoplan for patients with paroxysmal nocturnal hemoglobinuria and mild or moderate anemia (hemoglobin >/=10 g/dL) who had received eculizumab or were naive to complement inhibitors. PLoS One. 2024 Jul 29;19(7):e0306407. doi: 10.1371/journal.pone.0306407. eCollection 2024. PMID 39079163
- [Derived] Mulherin BP, Yeh M, Al-Adhami M, Dingli D. Normalization of Hemoglobin, Lactate Dehydrogenase, and Fatigue in Patients with Paroxysmal Nocturnal Hemoglobinuria Treated with Pegcetacoplan. Drugs R D. 2024 Jun;24(2):169-177. doi: 10.1007/s40268-024-00463-9. Epub 2024 May 10. PMID 38727860
- [Derived] Fishman J, Wilson K, Drzewiecka A, Pochopien M, Dingli D. The cost-effectiveness of pegcetacoplan in complement treatment-naive adults with paroxysmal nocturnal hemoglobinuria in the USA. J Comp Eff Res. 2023 Oct;12(10):e230055. doi: 10.57264/cer-2023-0055. Epub 2023 Sep 1. PMID 37655691
- [Derived] Wojciechowski P, Wdowiak M, Hakimi Z, Wilson K, Fishman J, Nazir J, Toumi M. Mapping the EORTC QLQ-C30 onto the EQ-5D-5L index for patients with paroxysmal nocturnal hemoglobinuria in France. J Comp Eff Res. 2023 May;12(5):e220178. doi: 10.57264/cer-2022-0178. Epub 2023 Apr 13. PMID 37052120
- [Derived] Wong RSM, Navarro-Cabrera JR, Comia NS, Goh YT, Idrobo H, Kongkabpan D, Gomez-Almaguer D, Al-Adhami M, Ajayi T, Alvarenga P, Savage J, Deschatelets P, Francois C, Grossi F, Dumagay T. Pegcetacoplan controls hemolysis in complement inhibitor-naive patients with paroxysmal nocturnal hemoglobinuria. Blood Adv. 2023 Jun 13;7(11):2468-2478. doi: 10.1182/bloodadvances.2022009129. PMID 36848639
- [Derived] Wong R, Fishman J, Wilson K, Yeh M, Al-Adhami M, Zion A, Yee CW, Huynh L, Duh MS. Comparative Effectiveness of Pegcetacoplan Versus Ravulizumab and Eculizumab in Complement Inhibitor-Naive Patients with Paroxysmal Nocturnal Hemoglobinuria: A Matching-Adjusted Indirect Comparison. Adv Ther. 2023 Apr;40(4):1571-1589. doi: 10.1007/s12325-023-02438-9. Epub 2023 Feb 7. PMID 36750531
- [Derived] Del Pozo Martin Y. 2021 ASH annual meeting. Lancet Haematol. 2022 Feb;9(2):e92-e93. doi: 10.1016/S2352-3026(21)00384-7. Epub 2021 Dec 16. No abstract available. PMID 34922648

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in subjects with paroxysmal nocturnal hemoglobinuria (PNH) at 22 investigational sites. The study consisted of a screening period (up to 4 weeks), followed by a randomized controlled period (RCP) (26 weeks). All subjects who completed RCP rolled over into a separate open-label, long-term extension study (APL2-307) or completed the safety follow-up (34 weeks).
Pre-assignment Details: A total of 68 subjects were screened. Of which, 53 subjects with PNH who met all of the inclusion criteria and none of the exclusion criteria were randomized in a 2:1 ratio either to receive pegcetacoplan or to remain on their current standard of care (SoC) in RCP.
Groups:
- Pegcetacoplan: Subjects were received subcutaneous (SC) infusion of pegcetacoplan 1080 milligram (mg) twice weekly or every 3 days up to end of the RCP (Week 26). Subjects were not allowed to receive treatment with other complement inhibitors.
- Standard of Care: Subjects continued to receive SoC treatment but were not allowed to receive treatment with a complement inhibitor unless they qualified for pegcetacoplan escape therapy.
Period: Overall Study
Arm/Group | Pegcetacoplan | Standard of Care
Started | 35 | 18
SoC to Pegcetacoplan (Escape Therapy) | 0 | 11
Completed | 33 | 17
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) set included all subjects assigned to treatment.
Groups:
- Pegcetacoplan: Subjects were received SC infusion of pegcetacoplan 1080 milligram (mg) twice weekly or every 3 days up to end of the RCP (Week 26). Subjects were not allowed to receive treatment with other complement inhibitors.
- Total: Total of all reporting groups
Arm/Group | Pegcetacoplan | Standard of Care | Total
Number analyzed (Participants) | 35 | 18 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (12.70) | 49.1 (15.64) | 44.5 (14.00)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 33 | 14 | 47
  >=65 and <75 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 24
  Male | 19 | 10 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 2 | 14
  Not Hispanic or Latino | 23 | 16 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 0 | 2
  American Indian or Alaska Native | 9 | 2 | 11
  Asian | 23 | 16 | 39
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Achieved Hemoglobin (Hb) Stabilization
Description: The Hb stabilization was defined as avoidance of a >1 gram per deciliter (g/dL) decrease in Hb concentration from Baseline in the absence of transfusion through Week 26.
Time Frame: From Baseline (Day 1) up to Week 26
Population: The ITT set included all subjects assigned to treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Pegcetacoplan: Subjects were received SC infusion of pegcetacoplan 1080 mg twice weekly or every 3 days up to end of the RCP (Week 26). Subjects were not allowed to receive treatment with other complement inhibitors.
Arm/Group | Pegcetacoplan | Standard of Care
Number analyzed (Participants) | 35 | 18
Participants | 30 | 0
Statistical Analysis 1: Comparison: Pegcetacoplan vs Standard of Care; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test is stratified by number of packed red blood cell (PRBC) within 12 months prior to screening (<4, ≥ 4) reported in electronic data capture (EDC) data; Difference = 0.7311, 95% CI 2-sided [0.572 to 0.8902]

2. Primary Outcome: Change From Baseline in Lactate Dehydrogenase (LDH) Concentration At Week 26
Description: The LDH concentration was analyzed using an analysis of covariance (ANCOVA) model with a last observation carried forward (LOCF) and a baseline observation carried forward (BOCF) approach for handling missing data. Baseline was defined as average of measurements prior to first dose of pegcetacoplan or on or prior to randomization of SoC. Post baseline missing values are imputed using multiple imputation method with Markov Chain Mont Carlo method.
Time Frame: Baseline (Day 1) and Week 26
Population: The ITT set included all subjects assigned to treatment.
Measure: Least Squares Mean (Standard Error); unit: Units/Liter (U/L)
Arm/Group | Pegcetacoplan | Standard of Care
Number analyzed (Participants) | 35 | 18
Units/Liter (U/L) | -1870.47 (100.971) | -400.09 (312.988)
Statistical Analysis 1: Comparison: Pegcetacoplan vs Standard of Care; Test type: Superiority; p < 0.0001, ANCOVA — p-value for Baseline, strata and treatment is from LS mean of proc mixed and proc mianalyze based on parameter estimates; LS mean difference = -1470.38, 95% CI 2-sided [-2113.44 to -827.32]

3. Secondary Outcome: Number of Subjects With an Hb Response in the Absence of Transfusions
Description: An Hb response was defined as a =>1 g/dL increase in Hb from baseline at Week 26.
Time Frame: Baseline and Week 26
Population: The ITT set included all subjects assigned to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan | Standard of Care
Number analyzed (Participants) | 35 | 18
Participants | 25 | 1
Statistical Analysis 1: Comparison: Pegcetacoplan vs Standard of Care; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test is stratified by number of PRBC within 12 months prior to screening (<4, ≥ 4) reported in EDC data; Difference = 0.5411, 95% CI 2-sided [0.339 to 0.7431]

4. Secondary Outcome: Change From Baseline in Absolute Reticulocyte Count (ARC) at Week 26
Description: Blood samples were collected via direct venipuncture at the specific time points to determine ARC. Baseline was defined as average of measurements prior to first dose of pegcetacoplan or on or prior to randomization of SoC. Post baseline missing values are imputed using multiple imputation method with Markov Chain Mont Carlo method.
Time Frame: Baseline and Week 26
Population: The ITT set included all subjects assigned to treatment.
Measure: Least Squares Mean (Standard Error); unit: 10^9 cells/L
Arm/Group | Pegcetacoplan | Standard of Care
Number analyzed (Participants) | 35 | 18
10^9 cells/L | -123.26 (9.164) | -19.44 (25.209)
Statistical Analysis 1: Comparison: Pegcetacoplan vs Standard of Care; Test type: Superiority; p = 0.0002, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference = -103.82, 95% CI 2-sided [-158.9 to -48.74]

5. Secondary Outcome: Change From Baseline in Hb Concentration at Week 26
Description: Baseline was defined as average of measurements prior to first dose of pegcetacoplan or on or prior to randomization of SoC. Post baseline missing values are imputed using multiple imputation method with Markov Chain Mont Carlo method.
Time Frame: Baseline and Week 26
Population: The ITT set included all subjects assigned to treatment.
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Pegcetacoplan | Standard of Care
Number analyzed (Participants) | 35 | 18
g/dL | 2.94 (0.383) | 0.27 (0.759)
Statistical Analysis 1: Comparison: Pegcetacoplan vs Standard of Care; Test type: Superiority; p = 0.0019, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference = 2.67, 95% CI 2-sided [0.99 to 4.35]

6. Secondary Outcome: Percentage of Subjects Who Received Transfusion or Decrease of Hb >2 g/dL From Baseline
Description: Transfusion refers to any transfusion of PRBC, leukocyte-depleted red blood cells (LDPRC), leukocyte poor packed red blood cell (LPRC), leukocyte poor blood (LPB) or whole blood.
Time Frame: At Week 26
Population: The ITT set included all subjects assigned to treatment.
Measure: Number; unit: percentage of subjects
Arm/Group | Pegcetacoplan | Standard of Care
Number analyzed (Participants) | 35 | 18
percentage of subjects | 11.4 | 100
Statistical Analysis 1: Comparison: Pegcetacoplan vs Standard of Care; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test is stratified by number of PRBC within 12 months prior to screening (<4, ≥4) reported in EDC data; Difference = -0.7505, 95% CI 2-sided [-0.9041 to -0.5969]

7. Secondary Outcome: Percentage of Subjects With Transfusion Avoidance
Description: Transfusion avoidance was defined as the percentage of subjects who did not require a transfusion during the RCP. Transfusion refers to any transfusion of PRBC, LDPRC, LPRC, LPB or whole blood.
Time Frame: At Week 26
Population: The ITT set included all subjects assigned to treatment.
Measure: Number; unit: percentage of subjects
Arm/Group | Pegcetacoplan | Standard of Care
Number analyzed (Participants) | 35 | 18
percentage of subjects | 91.4 | 5.6
Statistical Analysis 1: Comparison: Pegcetacoplan vs Standard of Care; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 6, analysis 1]; Difference = 0.7241, 95% CI 2-sided [0.5583 to 0.8899]

8. Secondary Outcome: Number of PRBC Units Transfused From Baseline Through Week 26
Description: The number of units of PRBC transfusions was estimated. In one transfusion subjects received one or more units.
Time Frame: Up to Week 26
Population: The ITT set included all subjects assigned to treatment.
Measure: Median (Full Range); unit: PRBC transfusions
Arm/Group | Pegcetacoplan | Standard of Care
Number analyzed (Participants) | 35 | 18
PRBC transfusions | 0.0 [0 to 19] | 3.0 [0 to 13]
Statistical Analysis 1: Comparison: Pegcetacoplan vs Standard of Care; Test type: Superiority; p < 0.0001, Wilcoxon Rank-Sum Test — Wilcoxon rank-sum test p-value for the comparison between treatments is based on median using stratified non-parametric analysis. The 95% confidence interval (CI) is constructed using Hodges-Lehmann Estimation of Location Shift; Median Difference (Net) = 3, 95% CI 2-sided [2 to 4]

9. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy- (FACIT-Fatigue) Scale Score at Week 26
Description: The FACIT-Fatigue Scale is a 13-item Likert scaled instrument that is self-administered by the subjects during clinic visits. Subjects were presented with 13 statements and asked to indicate their responses as it applied to the past 7 days. The 5 possible responses are "Not at all" (0), "A little bit" (1), "Somewhat" (2), "Quite a bit" (3), and "Very much" (4). With 13 statements, the total score has a range of 0 to 52. The higher score corresponded to a higher quality of life. Baseline is defined as average of measurements prior to first dose of pegcetacoplan or on or prior to randomization of SoC. Post baseline missing values are imputed using multiple imputation method with Markov Chain Mont Carlo method.
Time Frame: Baseline and Week 26
Population: The ITT set included all subjects assigned to treatment.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pegcetacoplan | Standard of Care
Number analyzed (Participants) | 35 | 18
scores on a scale | 7.78 (1.210) | 3.26 (2.113)
Statistical Analysis 1: Comparison: Pegcetacoplan vs Standard of Care; Test type: Superiority; p = 0.061, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference = 4.51, 95% CI 2-sided [-0.21 to 9.24]

10. Secondary Outcome: Percentage of Subjects With Hb Normalization Levels at Week 26
Description: Normalization of Hb levels defined as >= 1x LLN at Week 26 in the absence of transfusion. Transfusion refers to any transfusion of PRBC, LDPRC, LPRC, LPB or whole blood.
Time Frame: Baseline and Week 26
Population: The ITT set included all subjects assigned to treatment.
Measure: Number; unit: percentage of subjects
Arm/Group | Pegcetacoplan | Standard of Care
Number analyzed (Participants) | 35 | 18
percentage of subjects | 45.7 | 0
Statistical Analysis 1: Comparison: Pegcetacoplan vs Standard of Care; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Difference = 0.3645, 95% CI 2-sided [0.1648 to 0.5642]

11. Secondary Outcome: Percentage of Subjects With LDH Normalization at Week 26
Description: The LDH normalization was defined as LDH <= 1xupper limit of normal (ULN) of normal range at week 26 in the absence of transfusion. Transfusion refers to any transfusion of PRBC, LDPRC, LPPRC, LPRC, LPB or whole blood.
Time Frame: At Week 26
Population: The ITT set included all subjects assigned to treatment.
Measure: Number; unit: percentage of subjects
Arm/Group | Pegcetacoplan | Standard of Care
Number analyzed (Participants) | 35 | 18
percentage of subjects | 65.7 | 0
Statistical Analysis 1: Comparison: Pegcetacoplan vs Standard of Care; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference = 0.5592, 95% CI 2-sided [0.3682 to 0.7502]

12. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) 30-item Core Quality of Life Questionnaire (QLQ-C30) Scores at Week 26
Description: The EORTC QLQ-C30 questionnaire (version 3.0) consisted of 30 questions comprised of both multi-item scales and single-item measures to assess overall quality of life in subjects. Questions were designated by functional scales, symptom scales, and global subject QOL/overall perceived health status. For the first 28 questions the 4 possible responses are "Not at all' (1), 'A little' (2), 'Quite a bit' (3) and 'Very much' (4). For the remaining 2 questions the response is requested on a 7-point scale from 1 ('Very poor') to 7 ('Excellent'). Each scale has a range of 0% - 100%. A high scale score represents a higher response level. Baseline is defined as average of measurements prior to first dose of pegcetacoplan or on or prior to randomization of SoC. Post baseline missing values are imputed using multiple imputation method with Markov Chain Mont Carlo method.
Time Frame: Baseline and Week 26
Population: The ITT set included all subjects assigned to treatment.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pegcetacoplan | Standard of Care
Number analyzed (Participants) | 35 | 18
scores on a scale | 18.90 (2.909) | -2.85 (5.703)
Statistical Analysis 1: Comparison: Pegcetacoplan vs Standard of Care; Test type: Superiority; p = 0.0006, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference = 21.75, 95% CI 2-sided [9.35 to 34.16]

13. Secondary Outcome: Change From Baseline in Linear Analog Assessment (LASA) Scales Score at Week 26
Description: The LASA consisted of 3 items asking respondents to rate their perceived level of functioning. Specific domains include activity level, ability to carry out daily activities, and an item for overall QOL. Their level of functioning was reported on a 0-100 scale with 0 representing "As low as could be" and 100 representing "As high as could be".
Time Frame: Baseline and Week 26
Population: The ITT set included all subjects assigned to treatment.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pegcetacoplan | Standard of Care
Number analyzed (Participants) | 35 | 18
scores on a scale | 50.39 (9.062) | -5.39 (17.689)
Statistical Analysis 1: Comparison: Pegcetacoplan vs Standard of Care; Test type: Superiority; p = 0.005, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference = 55.79, 95% CI 2-sided [16.83 to 94.74]

14. Secondary Outcome: Percentage of Subjects With ARC Normalization
Description: Absolute reticulocyte count normalization is defined as ARC < 1x ULN of the gender-specific normal range at week 26 in the absence of transfusion. Subjects who received a transfusion or withdraw from study or escaped from SoC to pegcetacoplan treatment group or lost to follow up without providing efficacy data at Week 26 were classified as non-responders. Transfusion refers to any transfusion of PRBC, LDPRC, LPRC, LPB or whole blood.
Time Frame: At Week 26
Population: The ITT set included all subjects assigned to treatment.
Measure: Number; unit: percentage of subjects
Arm/Group | Pegcetacoplan | Standard of Care
Number analyzed (Participants) | 35 | 18
percentage of subjects | 60.0 | 5.6
Statistical Analysis 1: Comparison: Pegcetacoplan vs Standard of Care; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Difference = 0.4639, 95% CI 2-sided [0.2529 to 0.675]

15. Secondary Outcome: Number of Subjects With Failure of Hb Stabilization
Description: Hb stabilization is defined as avoidance of a >1 g/dL decrease in Hb levels from baseline through Week 26 in the absence of transfusion. Transfusion refers to any transfusion of PRBC, LDPRC, LPRC, LPB or whole blood.
Time Frame: Up to Week 26
Population: The ITT set included all subjects assigned to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan | Standard of Care
Number analyzed (Participants) | 35 | 18
Participants | 4 | 18
Statistical Analysis 1: Comparison: Pegcetacoplan vs Standard of Care; Test type: Superiority; p < 0.0001, Stratified Wilcoxon — Hazard ratio is based on cox proportional hazards model; Stratified Hazard Ratio = 0.02, 95% CI 2-sided [0.004 to 0.091]

16. Secondary Outcome: Time to First PRBC Transfusion
Description: Time to first-on-study PRBC transfusions during RCP were reported. Here NA indicates not estimable.
Time Frame: Up to Week 26
Population: The ITT set included all subjects assigned to treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pegcetacoplan | Standard of Care
Number analyzed (Participants) | 35 | 18
weeks | NA [NA to NA] — NA indicates that it was not possible to calculate a median and 95% confidence interval for time to first PRBC transfusion as fewer than 10% of subjects in the pegcetacoplan arm were transfused. | 7.000 [4.143 to 10.286]
Statistical Analysis 1: Comparison: Pegcetacoplan vs Standard of Care; Test type: Superiority; p < 0.0001, Stratified Wilcoxon; Stratified Hazard Ratio = 0.025, 95% CI 2-sided [0.005 to 0.121]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were reported from the first dose of study medication and for up to 8 weeks after the last dose of study medication, approximately 34 weeks.
Description: The safety set included all subjects who received at least 1 dose of pegcetacoplan and all subjects who were randomized to SoC. Overall Pegcetacoplan included 11 subjects who escaped from the SoC group to pegcetacoplan group.
Groups:
- Overall Pegcetacoplan: Subjects were received SC infusion of pegcetacoplan 1080 mg twice weekly or every 3 days up to end of the RCP (Week 26). Subjects were not allowed to receive treatment with other complement inhibitors. During the study, any subject assigned to the SoC reporting group (excluding complement inhibitors) who had an Hb concentration >=2 g/dL below baseline or who presented with a qualifying thromboembolic event secondary to PNH was offered early escape therapy with pegcetacoplan.
Arm/Group | Overall Pegcetacoplan | Standard of Care
All-Cause Mortality (participants affected / at risk) | 1/46 | 1/18
Serious Adverse Events (participants affected / at risk) | 6/46 | 3/18
Other Adverse Events (participants affected / at risk) | 35/46 | 12/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Pegcetacoplan (N=46) | Standard of Care (N=18)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dermoid cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Pegcetacoplan (N=46) | Standard of Care (N=18)
Pyrexia (General disorders) | 4 (4) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (2)
Malaise (General disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Viral infection (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (7) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (8) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (9) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 5 (10) | 0 (0)
Headache (Nervous system disorders) | 4 (9) | 0 (0)
Somnolence (Nervous system disorders) | 3 (3) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT04085601/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/01/NCT04085601/SAP_001.pdf